CLINICAL TRIAL: NCT02842528
Title: Study of Mental Flexibility and Inhibition Processes as Cognitive Vulnerability Markers of Alcohol Dependence
Brief Title: Cognitive Vulnerability Factors in Alcohol-dependence
Acronym: CoVAD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: PHRC-IR2006
Record Dates: First submitted 2016-06-27; First posted 2016-07-25 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-07

CONDITIONS: Alcoholism
MeSH Terms: conditions — Alcoholism | interventions — Wisconsin Card Sorting Test

ARMS (3):
- Alcohol-dependent patients (Experimental)
  Interventions: Behavioral: Diagnostic Interview for Genetic Studies; Behavioral: Family Informant Schedule and Criteria; Behavioral: Temperament and Character Inventory; Behavioral: Barratt Impulsiveness Scale; Behavioral: Wisconsin Card Sorting Test; Genetic: blood sample withdrawn
- First-degree relatives of alcohol-dependent probands (Active Comparator)
  Interventions: Behavioral: Diagnostic Interview for Genetic Studies; Behavioral: Family Informant Schedule and Criteria; Behavioral: Temperament and Character Inventory; Behavioral: Barratt Impulsiveness Scale; Behavioral: Wisconsin Card Sorting Test; Genetic: blood sample withdrawn
- Healthy Controls (Active Comparator)
  Interventions: Behavioral: Diagnostic Interview for Genetic Studies; Behavioral: Family Informant Schedule and Criteria; Behavioral: Temperament and Character Inventory; Behavioral: Barratt Impulsiveness Scale; Behavioral: Wisconsin Card Sorting Test; Genetic: blood sample withdrawn

INTERVENTIONS:
Behavioral: Diagnostic Interview for Genetic Studies
Behavioral: Family Informant Schedule and Criteria
Behavioral: Temperament and Character Inventory
Behavioral: Barratt Impulsiveness Scale
Behavioral: Wisconsin Card Sorting Test
Genetic: blood sample withdrawn

SUMMARY:
The purpose of this study is to specify the cognitive and genetic pattern associated with alcohol dependence. Results will help identifying more precisely vulnerability factors associated with this disorder.

DETAILED DESCRIPTION:
Alcohol dependence involves both environmental and genetic vulnerability factors. Although it has a rather high degree of heritability (estimates range between 40% and 60%), vulnerability to alcohol dependence is broadly recognised as a complex polygenic phenotype. To clarify the risk factors involved in alcohol dependence, attempts have been made to identify endophenotypes in alcohol dependent patients and their relatives. Endophenotypes are defined as heritable traits associated with an increased risk for developing a disorder; they must be found in probands and their unaffected relatives at a higher rate than in the general population and must be associated with a specific genetic pattern. In the present study the investigators investigate the cognitive performance of alcohol dependent patients in comparison with a group of adult non-alcoholic offspring of alcohol-dependent patients and a group of participants without family history of alcohol dependence. The investigators also explore the relation between familial density of alcoholism and cognitive performance, particularly mental flexibility and inhibition. Genetic analysis will also be conducted to investigate the relationship between cognitive performance and genetic patterns (single nucleotide polymorphisms).

ELIGIBILITY:
Inclusion Criteria:

Alcohol-dependent patients :

* Males or females, aged 18-65 years, with a diagnosis of alcohol dependence, according to the DSM-IV criteria
* Patients withdrawn from alcohol at least 2 weeks
* Native French speaker, able to read French and complete study evaluations
* Caucasian
* Able to provide informed written and verbal consent

First-degree relatives of alcohol-dependent probands :

* Males or females, aged 18-65 years
* Caucasian
* Native French speaker, able to read French and complete study evaluations
* Able to provide informed written and verbal consent

Healthy Controls :

* Males or females, aged 18-65 years
* Caucasian
* Native French speaker, able to read French and complete study evaluations
* Able to provide informed written and verbal consent

Exclusion Criteria:

Alcohol-dependent patients

* DSM-IV substance use disorder other than alcohol
* Severe chronic psychiatric disorders including Bipolar disorder and schizophrenia
* Mood episode diagnostic according to the DSM-IV criteria in the last six months
* A significant general medical illness, including neurological disorders
* A sensorial impairment uncorrected (visual and/or hearing)
* Individuals who are not covered by national health insurance

First-degree relatives of alcohol-dependent probands :

* Past or recent alcohol and/or drug abuse or dependence
* Severe chronic psychiatric disorders including Bipolar disorder and schizophrenia
* Mood episode diagnostic according to the DSM-IV criteria in the last six months
* A significant general medical illness, including neurological disorders
* Handling of psychotropics substances
* A sensorial impairment uncorrected (visual and/or hearing)
* Individuals who are not covered by national health insurance

Healthy Controls :

* A personal or first-degree-relative history of alcohol dependence
* Past or recent alcohol and/or drug abuse or dependence
* Total abstinence from alcohol
* Severe chronic psychiatric disorders including Bipolar disorder and schizophrenia
* Mood episode diagnostic according to the DSM-IV criteria in the last six months
* A significant general medical illness, including neurological disorders
* Handling of psychotropics substances
* A sensorial impairment uncorrected (visual and/or hearing)
* Individuals who are not covered by national health insurance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2007-09; Primary Completion 2009-03 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
questionnaire | Day 0
  comparison of questionnaires score for the 3 groups

SECONDARY OUTCOMES:
genetic polymorphism | Day 0

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Reims, Reims, France, France

REFERENCES:
- [Background] Gierski F, Hubsch B, Stefaniak N, Benzerouk F, Cuervo-Lombard C, Bera-Potelle C, Cohen R, Kahn JP, Limosin F. Executive functions in adult offspring of alcohol-dependent probands: toward a cognitive endophenotype? Alcohol Clin Exp Res. 2013 Jan;37 Suppl 1:E356-63. doi: 10.1111/j.1530-0277.2012.01903.x. Epub 2012 Dec 14. PMID 23240659
- [Background] Benzerouk F, Gierski F, Gorwood P, Ramoz N, Stefaniak N, Hubsch B, Kaladjian A, Limosin F. Brain-derived neurotrophic factor (BDNF) Val66Met polymorphism and its implication in executive functions in adult offspring of alcohol-dependent probands. Alcohol. 2013 Jun;47(4):271-4. doi: 10.1016/j.alcohol.2013.03.001. Epub 2013 Apr 10. PMID 23582695
- [Background] Raucher-Chene D, Gierski F, Hubsch B, Cuervo-Lombard CV, Bera-Potelle C, Cohen R, Kahn JP, Kaladjian A, Limosin F. Depression, anxiety and personality dimensions in female first-degree relatives of alcohol-dependent probands. Arch Womens Ment Health. 2012 Jun;15(3):229-32. doi: 10.1007/s00737-012-0271-5. Epub 2012 Mar 13. PMID 22411191
- [Background] Benzerouk F, Gierski F, Raucher-Chene D, Ramoz N, Gorwood P, Kaladjian A, Limosin F. Association study between reward dependence and a functional BDNF polymorphism in adult women offspring of alcohol-dependent probands. Psychiatr Genet. 2015 Oct;25(5):208-11. doi: 10.1097/YPG.0000000000000099. PMID 26204172